CLINICAL TRIAL: NCT02054026
Title: Impact Evaluation of the Reducing the Risk Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRP699102
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reducing the Risk (Experimental): An eight-lesson (approximately eight-hour) version of Reducing the Risk
  Interventions: Behavioral: Reducing the Risk
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Reducing the Risk
  Arms: Reducing the Risk

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an eight-hour version of Reducing the Risk on outcomes such as sexual initiation, condom and contraceptive use, number of sexual partners, and pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 9th grader
* Attends participating school

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2220 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sexual Initiation | 2-years post intervention

SECONDARY OUTCOMES:
Sexual Initiation | 1-year post intervention
Contraceptive use | 1-year post intervention
Contraceptive use | 2-years post intervention
Number of sexual partners | 1-year post intervention
Number of sexual partners | 2-years post intervention

OTHER OUTCOMES:
Attitudes towards healthy relationships and sexual activity | 1-year post intervention
Attitudes towards healthy relationships and sexual activity | 2-years post intervention
Knowledge of Sexually Transmitted Diseases | 1-year post intervention
Knowledge of Sexually Transmitted Diseases | 2-years post intervention
Career and Education Goals | 1-year post intervention
Career and Education Goals | 2-years post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, PhD, Study Director — Mathematica Policy Research
Locations (13):
- United States (13):
  - Bardstown High School, Bardstown, Kentucky
  - Warren Central High School, Bowling Green, Kentucky
  - Warren East High School, Bowling Green, Kentucky
  - Greenwood High School, Bowling Green, Kentucky
  - Central Hardin High School, Cecilia, Kentucky
  - Metcalfe County High School, Edmonton, Kentucky
  - Elizabethtown High School, Elizabethtown, Kentucky
  - Franklin-Simpson High School, Franklin, Kentucky
  - LaRue High School, Hodgenville, Kentucky
  - Marion County High School, Lebanon, Kentucky
  - North Hardin High School, Radcliff, Kentucky
  - Logan County High School, Russellville, Kentucky
  - Russellville Junior/Senior High School, Russellville, Kentucky